CLINICAL TRIAL: NCT00683787
Title: Multicenter Randomized Phase II Trial of Docetaxel With/Without VANDETANIB for Advanced Gastroesophageal Cancer
Brief Title: Docetaxel With or Without Vandetanib in Treating Patients With Metastatic Stomach Cancer or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000596150; RPCI-I-106207 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Active Comparator): Patients receive docetaxel IV once every 3 weeks.
  Interventions: Drug: docetaxel
- Arm II (Experimental): Patients receive docetaxel IV as in arm I and oral vandetanib (100 mg) once daily.
  Interventions: Drug: docetaxel; Drug: vandetanib
- Arm III (Experimental): Patients receive docetaxel IV as in arm I and oral vandetanib (300 mg) once daily.
  Interventions: Drug: docetaxel; Drug: vandetanib

INTERVENTIONS:
Drug: docetaxel — Given IV once every 3 weeks
Drug: vandetanib — Oral vandetanib once daily
  Arms: Arm II; Arm III

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether docetaxel is more effective when given together with or without vandetanib.

PURPOSE: This randomized phase II trial is studying docetaxel to see how well it works compared with docetaxel given together with vandetanib in treating patients with metastatic stomach cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the hypothesis that the addition of a targeted agent, such as vandetanib, to standard chemotherapy with docetaxel will result in incremental responses in patients with metastatic gastric or gastroesophageal junction cancer.

Secondary

* To assess progression-free survival and overall survival of patients treated with this regimen.
* To study the toxicity profile of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to clinical site. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive docetaxel IV once every 3 weeks.
* Arm II: Patients receive docetaxel IV as in arm I and oral vandetanib (100 mg) once daily.
* Arm III: Patients receive docetaxel IV as in arm I and oral vandetanib (300 mg) once daily.

In all arms, courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric adenocarcinoma or gastroesophageal junction cancer

  * Metastatic disease
* Measurable disease
* No symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Potassium ≥ 4.0 mEq/L (supplementation allowed) and ≤ the CTCAE grade 1 upper limit
* Magnesium normal (supplementation allowed) and ≤ the CTCAE grade 1 upper limit
* Calcium normal and corrected serum calcium ≤ the CTCAE grade 1 upper limit

  * In cases where the serum calcium is below the normal range, calcium (adjusted for albumin) normal OR ionized calcium normal
* ALT and AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 12 weeks after completion of study therapy
* Atrial fibrillation allowed if controlled by medication
* LVEF ≥ 45% by MUGA or ECHO

Exclusion criteria:

* Evidence of severe or uncontrolled systemic disease
* Any concurrent condition which makes it undesirable for the patient to participate in the trial or which would jeopardize study compliance, in the Investigator's opinion
* Uncontrolled infection
* Coagulopathy (including warfarin or anti-coagulant related) or bleeding disorder
* Peripheral neuropathy ≥ grade 2
* Clinically significant cardiac event, including myocardial infarction or New York Heart Association class II-IV heart disease within the past 3 months
* Presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia
* History of arrhythmia (i.e., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) OR asymptomatic sustained ventricular tachycardia
* History of QTc prolongation as a result of other medication that required discontinuation of that medication
* Congenital long QT syndrome or a first degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block
* QTc with Bazett's correction that is unmeasurable or ≥ 480 msec on screening ECG

  * If a patient has QTc ≥ 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart)
  * The average OTc from the three screening ECGs must be < 480 msec in order for the patient to be eligible for the study
* Hypertension not controlled by medical therapy (systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 100 mm Hg)
* Currently active diarrhea (≥ grade 2) that may affect the ability of the patient to absorb vandetanib
* Previous or current malignancies of other histologies within the past 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* At least 4 weeks since prior chemotherapy or radiotherapy
* No more than one prior chemotherapy regimen for metastatic disease

  * Prior adjuvant therapy, including chemoradiotherapy, allowed
* At least 2 weeks since prior palliative radiotherapy

  * Up to 3750 cGy palliative radiotherapy to the stomach allowed
* No prior therapy with docetaxel
* More than 30 days since prior investigational agents
* More than 4 weeks since prior and no concurrent or planned participation in another experimental drug study
* More than 4 weeks since prior major surgery and recovered
* More than 2 weeks since prior and no concurrent medication that may cause QTc prolongation or induce Torsades de Pointes
* No concurrent amiodarone
* No concurrent potent inducers of CYP3A4 function (e.g., rifampicin, rifabutin, phenytoin, carbamazepine, barbiturates, or Hypericum perforatum [St. John wort])
* No prior enrollment or randomization to treatment in the present study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Docetaxel: Patients receive docetaxel IV once every 3 weeks.
  docetaxel: Given IV once every 3 weeks
- Arm B: Docetaxel+VANDETANIB (100 mg): Patients receive docetaxel IV as in arm I and oral vandetanib (100 mg) once daily.
  docetaxel: Given IV once every 3 weeks
  vandetanib: Oral vandetanib once daily
- Arm C: Docetaxel+VANDETANIB (300 mg): Patients receive docetaxel IV as in arm I and oral vandetanib (300 mg) once daily.
  docetaxel: Given IV once every 3 weeks
  vandetanib: Oral vandetanib once daily
Period: Overall Study
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Started | 3 | 3 | 2
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 2
Not completed — Progression | 3 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg) | Total
Number analyzed (Participants) | 3 | 3 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.67 (7.64) | 67 (3.61) | 60 (8.49) | 61.38 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Time Frame: 1 year
Population: Due to the study's early termination and inadequate number of patients no statistical inference of the primary and secondary aims were carried forth.
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Progression-free Survival
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Toxicity
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Docetaxel | Arm B: Docetaxel+VANDETANIB (100 mg) | Arm C: Docetaxel+VANDETANIB (300 mg)
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel (N=3) | Arm B: Docetaxel+VANDETANIB (100 mg) (N=3) | Arm C: Docetaxel+VANDETANIB (300 mg) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel (N=3) | Arm B: Docetaxel+VANDETANIB (100 mg) (N=3) | Arm C: Docetaxel+VANDETANIB (300 mg) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 0 (0) | 2 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (7) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (7) | 2 (3) | 2 (5)
Mucosal inflammation (General disorders) | 2 (3) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blood alkaline phosphatase (Investigations) | 1 (1) | 2 (3) | 2 (2)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 1 (3) | 0 (0)
Electrocardiogram QT corrected interval (Investigations) | 0 (0) | 1 (1) | 1 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 1 (2)
Haemoglobin (Investigations) | 1 (1) | 1 (2) | 0 (0)
International normalised ratio (Investigations) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (7) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients no statistical inference of the primary and secondary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes